CLINICAL TRIAL: NCT02755519
Title: Case Detection and Confirmation, Subtype Classification of Patients With Primary Aldosteronism
Brief Title: Optimizing Diagnosis Of Primary Aldosteronism
Acronym: ODPA
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, M.D., PhD, Chongqing Medical University
Other Study IDs: ODPA 2016
Record Dates: First submitted 2016-04-08; First posted 2016-04-29 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Primary Aldosteronism
Keywords: primary aldosteronism; confirmatory test; hypertension
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Primary Aldosteronism: 1. Those with hypertension, and with or without hypoglycemia;
  2. Those with PAC/PRC≥42.95 pg·mL-1/µIU·mL-1
- Non-Primary Aldosteronism: 1. Those with Primary Hypertension;
  2. Those with adrenal diseases except for Primary Aldosteronism

SUMMARY:
To optimize the confirmatory tests for primary aldosteronism.

DETAILED DESCRIPTION:
In this study, the investigators aim to optimize the three confirmatory tests: salt loading, captopril challenge and fludrocortisone suppression, and to confirm a better choice of confirming testing for single or combined diagnosis of primary aldosteronism. Additionally, the investigators plan to collect blood and tissue samples of PA patients for genetic testing, and to proceed a long-term follow-up for further investigating the mechanism underlying PA and evaluating the cardio-cerebrovascular complications risk.

ELIGIBILITY:
Inclusion Criteria:

* With hypertension;
* With adrenal diseases

Exclusion Criteria:

* Pregnant or during lactation period;
* Under 18 yr;
* BMI ≤ 19 or ≥ 35
* With Cancer medical history
* Been through cardiovascular diseases in the past 3 months;
* Been through malignant arrhythmia, respiratory muscle paralysis or skeletal muscle paralysis caused by hypokalemia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group 1: Who was diagnosed with hypertension according to JNC standard and was considered with the possibility of primary aldosteronism.
  Group 2: Control Groups, one group for those without hypertension or with primary hypertension; the other group for those with adrenal diseases except for primary aldosteronism.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve (AUC) for Salt loading test | 1 week
  Salt loading test will be performed and compared to golden standard such as adrenal venous sampling (AVS) and biopsy results. The area under the curve (AUC) will be calculated.
AUC for captopril challenge test | 1 week
  Captopril challenge test will be performed and compared to golden standard such as AVS and biopsy results. AUC will be calculated.
AUC for fludrocortisone suppression test | 1 week
  Fludrocortisone suppression test will be performed and compared to golden standard such as AVS and biopsy results. AUC will be calculated.

SECONDARY OUTCOMES:
Incidence of cardiovascular diseases in Primary Aldosteronism | 3 years
  Follow-up for the risk of cardiovascular diseases, chronic kidney disease and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, M.D., PhD., Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Rossi GP, Belfiore A, Bernini G, Desideri G, Fabris B, Ferri C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Montemurro D, Palumbo G, Rizzoni D, Rossi E, Semplicini A, Agabiti-Rosei E, Pessina AC, Mantero F; PAPY Study Investigators. Prospective evaluation of the saline infusion test for excluding primary aldosteronism due to aldosterone-producing adenoma. J Hypertens. 2007 Jul;25(7):1433-42. doi: 10.1097/HJH.0b013e328126856e. PMID 17563566
- [Background] Ahmed AH, Cowley D, Wolley M, Gordon RD, Xu S, Taylor PJ, Stowasser M. Seated saline suppression testing for the diagnosis of primary aldosteronism: a preliminary study. J Clin Endocrinol Metab. 2014 Aug;99(8):2745-53. doi: 10.1210/jc.2014-1153. Epub 2014 Apr 24. PMID 24762111
- [Background] Li Y, Liu Y, Li J, Wang X, Yu Y. Sodium Infusion Test for Diagnosis of Primary Aldosteronism in Chinese Population. J Clin Endocrinol Metab. 2016 Jan;101(1):89-95. doi: 10.1210/jc.2015-2840. Epub 2015 Nov 13. PMID 26565948
- [Background] Nanba K, Tamanaha T, Nakao K, Kawashima ST, Usui T, Tagami T, Okuno H, Shimatsu A, Suzuki T, Naruse M. Confirmatory testing in primary aldosteronism. J Clin Endocrinol Metab. 2012 May;97(5):1688-94. doi: 10.1210/jc.2011-2504. Epub 2012 Mar 14. PMID 22419718
- [Background] Schirpenbach C, Seiler L, Maser-Gluth C, Rudiger F, Nickel C, Beuschlein F, Reincke M. Confirmatory testing in normokalaemic primary aldosteronism: the value of the saline infusion test and urinary aldosterone metabolites. Eur J Endocrinol. 2006 Jun;154(6):865-73. doi: 10.1530/eje.1.02164. PMID 16728547
- [Background] Agharazii M, Douville P, Grose JH, Lebel M. Captopril suppression versus salt loading in confirming primary aldosteronism. Hypertension. 2001 Jun;37(6):1440-3. doi: 10.1161/01.hyp.37.6.1440. PMID 11408392